CLINICAL TRIAL: NCT06661161
Title: Calibration of AlgoRithm for Detection of Cardiac Decompensation Via Parametric Objects
Brief Title: Calibration of AlgoRithm for Detection of Cardiac Decompensation Via Parametric Objects (CARDCOP)
Acronym: CARDCOP
Status: Not yet recruiting | Type: Observational
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Other Study IDs: 29BRC24.0222 - CARDCOP
Record Dates: First submitted 2024-09-30; First posted 2024-10-28 (Actual); Last update posted 2024-10-28 (Actual); Status verified 2024-10

CONDITIONS: Heart Failure - NYHA II - IV

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The goal of the study is to calibrate the algorithmic model of the TakeCoeur AI device to detect early heart failure decompensation in patients with heart failure, using physiological data (clinical) actively and passively collected through connected medical devices (watch, blood pressure monitor, and scale).

DETAILED DESCRIPTION:
In France, more than one million people suffer from chronic heart failure (HF) with an average age of 75 years. HF is a major public health issue, leading to 160,000 hospitalizations and 70,000 deaths each year, with an annual hospitalization cost estimated at €1.6 billion. Heart failure remains the third leading cause of cardiovascular mortality, with a 6 to 9 times higher risk of sudden cardiac death in HF patients compared to the general population.

After the age of 80, approximately 25% of heart failure patients die within three months of a decompensation episode, and nearly 40% within a year. Despite significant progress, the therapeutic management of patients remains complex, and hospitalizations are difficult to anticipate. It is even estimated that nearly 400,000 to 700,000 people with HF remain undiagnosed in France. Avoidable hospitalizations contribute to a deterioration in the quality of life for these patients and sometimes result in death.

Heart failure is a condition characterized by gradual worsening. Initially, the patient may be asymptomatic but progressively start to experience several, if not all, of the following symptoms: marked shortness of breath (dyspnea), edema, difficulty breathing when lying down (orthopnea), rapid weight gain, chronic fatigue, heart palpitations, and a drop in blood pressure upon standing. Monitoring the evolution of these symptoms is crucial to identifying the risk of heart failure decompensation and allowing for early and appropriate intervention to avoid hospitalization.

The progression of these symptoms can be tracked through the monitoring of physiological (clinical) variables such as weight, blood pressure, heart rate, and oxygen saturation. These are widely recognized parameters as indicators of health status and are frequently used in heart failure patient monitoring algorithms, as shown by systematic reviews.

Weight is one of the mandatory parameters to be collected according to HAS recommendations. The American Heart Failure Association (HFSA) and the guidelines of the European Society of Cardiology (ESC) also recommend daily weight monitoring. Blood pressure is also among the recommended clinical symptoms to monitor, as it is a precursor sign of heart failure decompensation.

The four warning signals-shortness of breath, rapid weight gain, lower limb edema, and fatigue (EPOF)-must be monitored, especially after the age of 60, to promote early diagnosis and prevent hospitalizations.

Resting and exercise heart rates can predict the risk of cardiovascular disease. A high resting heart rate is associated with an increased risk of coronary heart disease and all-cause mortality and is also considered a predictive factor for decompensation in HF patients. Respiratory rate has been found to be significantly lower in patients with heart failure decompensation. However, physical activity is linked to better cardiovascular health and reduced mortality . Recommended by the American Heart Association (AHA) as one of the "8 Simple Measures for a Healthy Life", physical activity helps promote heart health.

Continuous and real-time collection of all these physiological (clinical) parameters in heart failure patients at risk of decompensation could improve patient follow-up and help predict the risk of acute heart failure decompensation. Indeed, a better understanding of these parameters, their variations, and their correlations would allow for better characterization of heart failure patients and early identification of decompensation.

This study aims to identify predictive factors of heart failure decompensation to develop and train an early detection algorithm that will be used in telemonitoring after the algorithm's calibration. To collect this data stream, heart failure patients will be equipped with three connected devices (watch, scale, blood pressure monitor) linked to the TakeCoeur AI device. The early detection algorithm for heart failure decompensation will be built based on variations in the physiological parameters collected and the occurrence of heart failure decompensation during the study period.

The patient's clinical data will be collected by the cardiologist at inclusion, and the physiological parameters will be passively and actively collected through connected devices. A baseline for each patient will be established at inclusion, reflecting their initial status. Throughout the study, any deviation or variation from this baseline will be detected. In case of a heart failure decompensation, a link between this decompensation and the variations in digitally collected parameters will be established.

The investigators hypothesize that the early detection of heart failure decompensation by the TakeCoeur AI device will align with the actual occurrence of heart failure decompensation, as recorded through healthcare utilization during this study, with good sensitivity and a low rate of false negatives.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Patient diagnosed with chronic heart failure, confirmed by a cardiologist/cardio-geriatrician (regardless of the type and etiology of the disease), meeting at least one of the following two conditions:
* Hospitalization in the past 12 months for a heart failure exacerbation.
* NYHA class II to IV (New York Heart Association) at the time of inclusion, with elevated natriuretic peptide levels (BNP > 100 pg/mL or NT-proBNP > 1000 pg/mL).
* French speaking patient
* Patient equipped with a smartphone, computer, or tablet with internet/cellular access (of with the help of a caregiver)
* Patient affiliated with a social security scheme

Exclusion Criteria:

* Patient undergoing dialysis for renal failure
* Patient who has received or is scheduled to receive a heart transplant or circulatory assistance within the next 12 months
* Patient with a left ventricular ejection fraction ≥ 50% (for non-diastolic heart failure)
* Obese patient with a body mass index ≥ 40 kg/m²
* Patient with severe aortic stenosis who is contraindicated for surgery or TAVI
* Patient with a life expectancy of < 1 year due to a condition other than heart failure (cancer, cirrhosis, respiratory failure, etc.)
* Patient already benefiting from a telemonitoring device
* Physical or psychological inability (dementia, schizophrenia, substance-related disorder) of the patient or caregiver to use the digital data collection device, as judged by the physician
* Patient refusal to allow the transmission of the data necessary for monitoring the effective use of the device and obtaining individualized or national real-world usage results
* Patient under guardianship, curatorship, or any other administrative or judicial measure restricting rights and freedoms
* Patient unable to wear the watch for the duration of the study due to skin conditions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participation in the study will be offered to any patient consulting a cardiologist/cardio-geriatrician at one of the participating centers who meets the inclusion criteria and non inclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 640 (Estimated)
Dates: Start 2024-11 (Estimated); Primary Completion 2025-11 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Concordance between the detection of heart failure decompensation by the TakeCoeur AI device and the occurrence of heart failure decompensation | From enrollment to the end of the 6-month follow-up period.
  calibrate the algorithmic model of the TakeCoeur IA device for early detection of cardiac decompensation in patients suffering from heart failure.

SECONDARY OUTCOMES:
Evaluate the time (in days) to anticipate cardiac decompensation | From enrollment to the end of the 6-month follow-up period.
  time to predict (in days) the risk of cardiac decompensation
Evaluate the compliance of patients with heart failure to the Takecoeur IA device and its connected collection accessories | From enrollment to the end of the 6-month follow-up period.
  - Monthly questionnaire (scale 0 to 4 for edema and shortness of breath) completion rate defined by the following formula: (number of completed questionnaires / total number of questionnaires to be completed) x 100

CONTACTS AND LOCATIONS:
Locations (3):
- France (3):
  - Chu Brest, Brest
  - CH Morlaix, Morlaix
  - CH Vannes, Vannes

IPD SHARING:
Plan to Share IPD: Yes
All collected data that underlie results in a publication
Supporting Information: Study Protocol
Time Frame: Data will be available beginning three years and ending fifteen years following the final study report completion
Access Criteria: Data access requests will be reviewed by the internal committee of Brest UH. Requestors will be required to sign and complete a data access agreement